CLINICAL TRIAL: NCT01777737
Title: Pilot Study Phase III to Evaluate the Efficacy and Safety of Trimethoprim-sulfamethoxazole in the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Study to Test the Validity of the Treatment of Idiopathic Pulmonary Fibrosis With Cotrimoxazole
Acronym: TriSulfa-FPI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Changes in standards of care
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TriSulfa-FPI-1
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Trimethoprim-sulfamethoxazole; Pneumocystis jiroveci
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cotrimoxazole (Experimental): Sulfamethoxazole 400 mg. + trimethoprim 80 mg. weight-adjusted
  Interventions: Drug: Cotrimoxazole
- Placebo (Placebo Comparator): Identical capsules to cotrimoxazole
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cotrimoxazole — 24 weeks of treatment
  Arms: Cotrimoxazole
Drug: Placebo — Identical capsules to cotrimoxazole
  Other Names: Placebo with identical physical appearance
  Arms: Placebo

SUMMARY:
First study to test the validity of the treatment of idiopathic pulmonary fibrosis, which causes inflammation and fibrosis (scarring) of the lung tissue, with cotrimoxazole.

Cotrimoxazole may improve the clinical course of the disease through eradication of Pneumocystis jiroveci colonization and other mechanisms as inhibiting the activation of alveolar macrophages and producing alterations in the surfactant system which favours the persistent activation of the inflammatory response and the development of pulmonary fibrosis.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a chronic lung disease that is clinically manifested by the appearance of effort dyspnea and impaired lung function.

The natural history of the disease is poorly understood and there is no clear consensus as to the most appropriate markers for predicting patient outcome.

This pilot controlled trial aims to test the efficacy and safety of cotrimoxazole in the treatment of IPF. This novel therapeutic strategy, with very encouraging preliminary data is based on its pathophysiological basis, primarily related to the elimination of Pneumocystis colonization. That elimination, could serve as a potent weapon for reducing morbidity and mortality and the cost associated with this devastating disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient, regardless of gender, aged 18 to 80 years.
* Well-established diagnostic criteria of the Idiopathic Pulmonary Fibrosis (IPF) as ATA/ERS/JRS/ALAT 2011.
* Ability to obtain a sample of sputum or oropharyngeal washing.
* Forced Vital Capacity (FVC) above 50% from the theoretical value expected.
* Patient compliance or legal guardian to participate in this study by signing the informed consent.

Exclusion Criteria:

* Allergy / hypersensitivity or known gastrointestinal intolerance to cotrimoxazole.
* Use of immunosuppressants or corticosteroids in the previous 90 days at baseline.
* Exacerbation of IPF and / or pneumonia in the 90 days prior to baseline.
* Presence of autoimmune diseases or asthma.
* Patients with other significant diseases other than IPF. It is considered significant disease any disease or condition that, in the investigator's opinion, may jeopardize the patient's health participating in the study or influence the results of the study or the patient's ability to participate in the study.
* Pregnant or lactating or of childbearing potential not using medically approved contraceptive methods at least three months before or during trial.
* Participation in another trial with an investigational drug within 30 days or six half-lives (the larger of the two) above the baseline.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of oral cotrimoxazole versus placebo in idiopathic pulmonary fibrosis (IPF). | 24 weeks
  Decline of the FVC ≥ 5% at 24 weeks and / or hospitalization for respiratory causes.

SECONDARY OUTCOMES:
Evaluate the safety of oral cotrimoxazole versus placebo in IPF. | At 24 weeks
  * Time to progression
  * Any cause of hospitalization
  * Overall mortality
  * Incidence and severity of adverse events.
Evaluate the effect of cotrimoxazole on the natural history of Pneumocystis colonization in patients with IPF. | 24 weeks
  - Molecular diagnosis of colonization by Pneumocystis jiroveci.
Identify the effects of cotrimoxazole systemic level of inflammatory activity in patients with IPF. | At 24 weeks
  * Acute exacerbation of IPF
  * Scales of dyspnea
  * Reduction > 50% in the values of different proinflammatory cytokines
  * Reduction > 50% in the values of surfactant proteins.
  * Reduction > 50% in the values of chemokine CCL-18.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío/ Instituto de Biomedicina de Sevilla, Seville, Spain